CLINICAL TRIAL: NCT03166995
Title: Study of the Effect of a Postural Exercise Program in Women With Fibromyalgia: a Randomized Clinical Trial
Brief Title: Postural Exercises in Women With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Marta Inglés de la Torre, Principal investigator, University of Valencia
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: H1484818368873
Record Dates: First submitted 2017-05-23; First posted 2017-05-25 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia,postural exercises
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1 (Experimental): Low impact aerobic exercise group. 1hour, twice a week
  Interventions: Other: Low impact aerobic exercise
- Experimental group 2 (Experimental): Postural exercises group. 1hour, twice a week
  Interventions: Other: Postural exercises
- Control propriocepcion (No Intervention): No exercise, just proprioceptive control.

INTERVENTIONS:
Other: Low impact aerobic exercise — The intervention will consist of working the muscles that are most affected by FMS through group exercises, which will be dynamic, fluid and aimed at improving functionality. Each session will consist of 60 minutes and will be divided into three parts: warm up (15 minutes); games, group dynamics and aerobics (30 minutes); and cool down with stretching for 15 minutes.
  Arms: Experimental group 1
Other: Postural exercises — The intervention will consist of performing postural exercises in prone, supine, sitting and standing position, as well as in quadrupedia. Each session will consist of 60 minutes and will be divided into three parts: warm up (15 minutes); postural exercises (30 minutes); and cool down with stretching for 15 minutes.
  Arms: Experimental group 2

SUMMARY:
In the current study, the investigators aimed to study:

* The proprioception status of patients with FMS.
* The effectiveness of a postural exercise program in women with fibromyalgia for 8 weeks (2 sessions per week), compared to a low impact aerobic exercise program on different parameters, such as proprioception, balance, muscle strength, flexibility and joint range.

DETAILED DESCRIPTION:
Fibromyalgia syndrome (FMS) is a multisystemic disease, characterized by generalized chronic musculoskeletal pain. In addition, it is usually accompanied by fatigue, sleep disorders, morning stiffness, cognitive disorders, depression, anxiety and stress. Other common symptoms are back pain, headaches, irritable bowel, balance problems and deterioration of physical function.

It constitutes the second most common rheumatic 36 disorder after osteoarthritis, with a prevalence of 2.9% in Europe and a fivefold times greater incidence among women than men.

Patients with FMS have pain at specific pressure points known as "tender points", with increased sensitivity to painful stimuli (hyperalgesia) and a decreased pain threshold (allodynia), in the absence of abnormalities in the biological or imaging tests. These tender points constitute the basis of the most sensitive and specific criteria for the diagnosis of the disease, this is, the criteria of the American College of Rheumatology. Accordingly, women presenting at least 11 of 18 tender points are diagnosed with FMS.

The etiology of FMS remains unclear. However, the generalized hyperalgesia, widespread pain and spontaneous pain in FMS have been related to central changes, and many studies support a major role for central sensitization in the generation of the symptoms of FMS.

Since it is a chronic disease, the care of this type of patients represents a significant economic burden. They have great health care resource requirements in both direct medical care and indirect costs of staff absenteeism. For these reasons, it is considered a major problem with a great impact on the health system, and therefore more and more studies are being developed with the aim of better understanding the pathophysiology of this disease.

In general, the goal of the treatment should be to improve function. In this regard, some studies have demonstrated the efficacy of low-cost therapeutic measures, such as physical exercise programs, to improve FMS symptoms. Physical exercise has a direct effect on pain, joint and muscle stiffness, generalized sensitivity fatigue, cognitive function. Since there is no standard program, it is difficult to determine which exercise modality is most effective on FMS. Most studies focus on low-impact aerobic exercise performed between 60-70% of maximal heart rate two to three times a week.

On the other hand, it has been proposed that motor control problems, due mainly to an alteration of the central and peripheral system, are associated with muscle strength loss, motor or sensory deficits and suboptimal muscle coordination. The lack of balance may also be due to a disturbance in the perception or interpretation of auditory- vestibular signals. Therefore, postural stability training is recommended to stimulate the neuromuscular system and develop proprioceptive capacity aimed at improving motor control and postural balance among these patients. In this regard, it is important to note that FMS is associated with postural control and balance impairments, the latter being one of the 10 most debilitating symptoms, with a prevalence of 45%.

In the current study, the investigators aimed to study:

* The proprioception status of patients with FMS.
* The effectiveness of a postural exercise program in women with fibromyalgia for 8 weeks (2 sessions per week), compared to a low impact aerobic exercise program on different parameters, such as proprioception, balance, muscle strength, flexibility and joint range.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 30 and 65 years.
* Meeting ACR 2010 criteria for FMS.

Exclusion Criteria:

* Medical contraindication for physical activity.
* Deafness or limited hearing.
* Vestibular disorders that compromise balance.
* Low vision or blindness.
* Psychotic disorder or cognitive impairment.
* Decompensation or changes in medication.
* Surgical interventions in the last six months.
* Rheumatic disease.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-12-29 (Actual)

PRIMARY OUTCOMES:
Proprioception | 8 weeks
  Proprioception will be evaluated at baseline and at the end of the study possible differences between women with fibromyalgia and healthy women using an isokinetic device (BIODEX MULTI-JOINT SYSTEM - PRO). The following movements were analized: knee (flexion, extension), hip (flexion, extension, abduction, adduction), ankle (flexion, extension), shoulder (flexion, extension). Joint position sense for knee extension and shoulder flexion will be also performed.

SECONDARY OUTCOMES:
Balance | 8 weeks
  Evaluated by the Berg Balance Scale. This consists of 14 items, in which static and dynamic balance is assessed. Subjects are asked to perform balance related tasks of varying difficulties (from standing up from a sitting position to monopedal standing). According to the ability to carry out the assessed activity, each task is scored on a 5-point scale (0= lowest level of function, 4= highest level of function). The final measure is the sum of all the scores (maximum=56 points) and higher scores are indicative of greater functional balance. This test has shown excellent intra-rater reliability (ICC = 0.97) and test-retest reliability (ICC = 0.91).
Handgrip strength | 8 weeks
  Grip strength will be measured by a Jamar Analogue Hand Dynamometer with participants seated, their elbow by their side and flexed to right angles, and a neutral wrist position. Subjects were verbally encouraged to produce their maximal grip strength (MGS). Three trials were recorded, consisting of a 3-second maximal contraction, with a 30-second rest period between each trial. The maximal value of the three reproducible trials for each hand was retained for analyses.
Joint range of motion | 8 weeks
  Ranges of movement of different joints were evaluated by a goniometer and an inclinometer: Shoulder (flexion, extension, abduction, adduction, internal and external rotation), hip (flexion, extension, abduction, adduction, internal and external rotation), knee (flexion and extension), ankle (flexion, extension, abduction, adduction, internal rotation and external rotation), cervical spine (flexion, extension, rotations and inclinations). For the measurements, subjects were in underwear or wore comfortable clothes.
Pain | 8 weeks
  Evaluated by the McGill Pain Questionnaire (MPQ). The MPQ includes 4 main measures:
  1. Pain location. On a drawing of the human body with both anterior and posterior sides, participants indicate the areas of their bodies that have pain. The number of pain sites is summed as in indicator of the sensory pain dimension.
  2. Pain intensity. From a list of 6 words, the patient selects the one best word describing the intensity of pain: 0 = none, 1= mild, 2 = discomforting, 3 = distressing, 4 = horrible and 5 = excruciating.
  3. Pain quality. Participants respond to the question, "What does your pain feel like?" by selecting from 78 descriptors in 20 subclasses. The quantitative data is summed to form the Pain Rating Index (PRI) (score 0 no pain- 78 worst possible pain).
  4. Pain pattern. Participants respond to the question, "How does your pain change with time?" by selecting from 9 words.
Leisure Time Physical Activity | 8 weeks
  Evaluated by the Leisure Time Physical Activity Instrument (LTPAI). It is an instrument assessing the amount of physical activity performed during a typical week. The physical activities are divided into three categories: light, moderate, and heavy activities. The LTPAI total score is the sum of hours in all three categories.
Impact on quality of life | 8 weeks
  Evaluated by the Fibromyalgia Impact Questionnaire (FIQ). This is a multidimensional self-administered questionnaire with 10 items that evaluates the status of the patient the week before the test is completed, and it assesses the aspects that tend to be more affected in people with FMS. The first item contains 10 sub-items, ranging from four points (from 0= always to 3 = never) and assesses the patient's functional capacity in activities of daily living. The second and third items refer to days of the week and the rest are visual analog scales from 0 to 10. The score ranges from 0 to 100, where 0 represents the maximal functional capacity quality of life and 100 the minimum. This scale was validated in its Spanish version by Salgueiro and García-Leiva in 2013, and it showed an excellent internal consistency (Cronbach's alpha = 0.95).
Anxiety and Depression | 8 weeks
  Assessed by the Hospital Anxiety and Depression Scale (HADS). This is a valid and reliable self-rating scale with 14 items that measures anxiety and depression (7 of the items relate to anxiety and 7 relate to depression). Each item is answered by the patient on a four point (0-3) response category so the possible scores range from 0 to 21 for anxiety and 0 to 21 for depression, with scores categorized as follows: normal 0-7, mild 8-10, moderate 11-14, and severe 15-21. Scores for the entire scale (emotional distress) range from 0 to 42, with higher scores indicating more distress.
Fatigue | 8 weeks
  Fatigue Severity Scale (FSS). The FSS is a self-administered questionnaire with 9 items (questions) investigating the severity of fatigue in different situations during the past week. Grading of each item ranges from 1 to 7, where 1 indicates strong disagreement and 7 strong agreement, and the final score represents the mean value of the 9 items.
Sleep disorders | 8 weeks
  Evaluated by the Pittsburgh Sleep Quality Index (PSQI). It is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Inglés, PhD, Principal Investigator — Faculty of Physiotherapy. University of Valencia
Locations (1):
- Faculty of Physiotherapy, University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No